CLINICAL TRIAL: NCT00822835
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ILV-095 Administered Subcutaneously to Healthy Subjects
Brief Title: Study Evaluating Single Doses of ILV-095 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 3226K1-1000
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ILV-095 (Active Comparator): 6 SC single dose injections
  Interventions: Biological: ILV-095
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ILV-095
  Arms: ILV-095
Biological: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single doses of ILV-095 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women of non-childbearing potential ages 18 to 50 years old.
2. Body mass index (BMI) in the range of 18 to 32 kg/m2 and body weight greater than or equal to50 kg.
3. Healthy as determined by the investigator on the basis of screening evaluations.
4. Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.
5. Have a high probability for compliance with and completion of the study.

Exclusion Criteria:

1. Presence or history of any disorder that may prevent the successful completion of the study.
2. Any subject who had orthopedic surgery within 12 weeks of the screening visit or has planned (elective) orthopedic surgery within 12 weeks of study drug administration.
3. Acute disease state (eg, nausea, vomiting, fever, active infection, or diarrhea) within 7 days before enrollment.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be evaluated from adverse events, physical examinations, vital sign measurements, cardiac rhythm monitoring, 12-lead ECGs, and clinical laboratory test results. | 3 weeks per group

SECONDARY OUTCOMES:
Pharmacokinetic parameters | 3 weeks per group

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Philadelphia, Pennsylvania, United States